CLINICAL TRIAL: NCT03091751
Title: Efficacy and Safety of Factor IX (FIX) Contained in AlphaNine® and Its Pharmacokinetic Comparison With BeneFIX® in Patients With Severe Hereditary Haemophilia B
Brief Title: Efficacy and Safety of AlphaNine Versus BeneFIX in Patients With Severe Hereditary Haemophilia B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG-404-1
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Results first posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Hemophilia B
Keywords: Factor IX (FIX)
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | US Export: Yes

ARMS (1):
- BeneFIX (Experimental): BeneFIX is a recombinant FIX provided in a vial containing 100 IU/mL lyophilized nonacog alfa accompanied with solvent for reconstitution and injection.
  Interventions: Drug: BeneFIX

INTERVENTIONS:
Drug: BeneFIX — BeneFIX is a recombinant FIX that contains nonacog alfa, reconstituted in solvent and administered as a single dose of 65-75 IU/kg.
  Other Names: recombinant coagulation factor IX

SUMMARY:
The goal of this non-randomized, multi-center study in subjects with severe hereditary haemophilia B was to determine and compare the pharmacokinetic and safety profiles of BeneFIX in subjects having had 2 prior pharmacokinetic assessments with AlphaNine.

DETAILED DESCRIPTION:
Two pharmacokinetic assessments (studies) were carried out in the same subjects during a previous clinical trial. The first pharmacokinetic study (PK1) was performed after a single dose of AlphaNine. The second pharmacokinetic study (PK2) was performed following 26 Weeks of AlphaNine treatment after PK1. To compare AlphaNine with BeneFIX, a third pharmacokinetic study (PK3) (current study) was performed after a single dose of BeneFIX administered following a 7- to 15-day wash-out period.

The main objective of the PK3 study was to assess the pharmacokinetic profile of BeneFIX and compare to the pharmacokinetic profile of AlphaNine from the PK2 study.

ELIGIBILITY:
Key Inclusion Criteria:

* Participated in the previous study "Efficacy and safety of factor IX (FIX) contained in Alphananine in patients with severe hereditary haemophilia B":
* Congenital deficiency in Factor IX (FIX)
* FIX residual activity of ≤2% of normal
* Had required FIX-containing products in the past and in clinical records that were collected data to assess a reliable estimation of at least 150 treatment exposure days to previous products
* Was able to receive treatment for more than 10 days for a 6-month period

Key Exclusion Criteria:

* Received a dose of FIX in the 7 days prior to the infusion
* FIX inhibitor level of >0.5 Bethesda units (BU) or clinically relevant presence in the past (≥5 BU)
* Active bleeding at the moment of infusion
* Had a known allergic reaction to any BeneFIX component
* Exhibited symptoms of any intercurrent infection (ie, fever, chills, nausea) at the time of the first infusion
* Had any disease that might affect the distribution or metabolism of FIX and which could affect interpretation of the study (such as non-controlled diabetes mellitus)
* Had non-controlled arterial hypertension
* Had abnormal renal function (creatinine >1.5 mg/dL)
* Had documented liver cirrhosis or any hepatic disorder with alanine aminotransferase (ALT) levels 2.5x upper limit of normal (ULN )
* Prevision to be concomitantly treated with other FIX-containing products
* Had conditions that might affect subject compliance (survival-limiting [in 2 year time] diseases, alcohol or other drug abuse, etc.)
* Unable to provide a storage plasma sample before the first dose of BeneFIX

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Bulgaria (3):
  - Medical University Pleven, Pleven
  - National Center of Haematology, Sofia
  - Medical University, University Hospital "Sveta Marina",, Varna

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BeneFIX
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Thirteen subjects with 2 prior pharmacokinetic assessments with AlphaNine (PK1, PK2) had a third PK assessment with BeneFIX (PK3). Nine subjects had PK3 analysis with BeneFIX as part of a previous study. In total, 22 subjects treated with BeneFIX (PK3) were analyzed jointly and compared to 25 subjects treated with AlphaNine (PK2).
Arm/Group | BeneFIX
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference of Area Under the Curve (AUC): BeneFIX Compared to AlphaNine
Description: BeneFIX pharmacokinetic parameter of area under the curve (AUC 0-inf) was assessed and compared to the AlphaNine pharmacokinetic parameter (PK2 study).
Time Frame: Baseline (prior to the infusion), and at 15 and 30 minutes, 1, 3, 6, 9, 24, 48, 72, and 74 hours following a single dose infusion of BeneFIX administered following a 7 to 15 day wash-out period.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: IU x hour/dL
Arm/Group | BeneFIX
Number analyzed (Participants) | 22
IU x hour/dL | 10.41 (563.081)
Statistical Analysis 1: Comparison: BeneFIX; Test type: Other; p = 0.77, t-test, 1 sided; Mean Difference (Final Values) = 10.41, 95% CI 2-sided [-224.88 to 245.70]

2. Primary Outcome: Mean Difference of In Vivo Recovery: BeneFIX Compared to AlphaNine
Description: BeneFIX pharmacokinetic parameter of in vivo recovery was assessed and compared to the AlphaNine pharmacokinetic parameter (PK2 Study).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: kg/dL
Arm/Group | BeneFIX
Number analyzed (Participants) | 22
kg/dL | 0.3068 (0.37505)
Statistical Analysis 1: Comparison: BeneFIX; Test type: Other; p = 0.002, t-test, 1 sided; Mean Difference (Final Values) = 0.3068, 95% CI 2-sided [0.1501 to 0.4635]

3. Primary Outcome: Mean Difference of Terminal Half-Life: BeneFIX Compared to AlphaNine
Description: BeneFIX pharmacokinetic parameter of terminal half-life was assessed and compared to the AlphaNine pharmacokinetic parameter (PK2 Study).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BeneFIX
Number analyzed (Participants) | 22
hours | -3.3 (13.48)
Statistical Analysis 1: Comparison: BeneFIX; Test type: Other; p = 0.30, t-test, 1 sided; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-8.9 to 2.3]

4. Primary Outcome: Mean Difference of Clearance: BeneFIX Compared to AlphaNine
Description: BeneFIX pharmacokinetic parameter of clearance was assessed and compared to the AlphaNine pharmacokinetic parameter (PK2 Study).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mL/min x kg
Arm/Group | BeneFIX
Number analyzed (Participants) | 22
mL/min x kg | -0.0058 (0.0145)
Statistical Analysis 1: Comparison: BeneFIX; Test type: Other; p = 0.16, t-test, 1 sided; Mean Difference (Final Values) = -0.0058, 95% CI 2-sided [-0.0119 to 0.0003]

5. Primary Outcome: Mean Difference of Mean Residence Time (MRT): BeneFIX Compared to AlphaNine
Description: BeneFIX pharmacokinetic parameter of mean residence time (MRT 0-inf) was assessed and compared to the AlphaNine pharmacokinetic parameter (PK2 Study).
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BeneFIX
Number analyzed (Participants) | 22
hours | -7.609 (13.7121)
Statistical Analysis 1: Comparison: BeneFIX; Test type: Other; p = 0.02, t-test, 1 sided; Mean Difference (Final Values) = -7.609, 95% CI 2-sided [-13.344 to -1.879]

ADVERSE EVENTS:
Time Frame: Adverse events produced during and after treatment administration were recorded.
Arm/Group | BeneFIX
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the study, after providing Sponsor 30 days' notice prior to submitting a manuscript or other materials related to the study to any outside party. At Sponsor's request, site will remove any confidential information (other than study results) and site will, upon Sponsor's request, delay publication or presentation for a period of up to 120 days to allow Sponsor to protect its interests in any Sponsor interventions.